CLINICAL TRIAL: NCT06905054
Title: Peroxisome Proliferator-Activated Receptor Agonists to Prevent Primary Sclerosing Cholangitis Recurrence After Liver Transplantation
Brief Title: Pharmacologic Approaches to Preventing Primary Sclerosing Cholangitis Recurrence After Liver Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Channa R Jayasekera, MD, MSc, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-007598
Record Dates: First submitted 2025-02-28; First posted 2025-04-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Primary Sclerosing Cholangitis; Liver Transplant, Complications; PSC; Biliary Strictures
Keywords: primary sclerosing cholangitis; recurrent primary sclerosing cholangitis; liver transplant complication; fenofibrate; fibrate; PPAR agonist; peroxisome proliferated activated receptor agonist
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Fenofibrate; Pharmaceutical Preparations; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Individuals who underwent liver transplantation for primary sclerosing cholangitis 1-7 years before study initiation, and meeting study criteria, will receive fenofibrate 160mg oral daily for 36 months
  Participants will undergo the following serum assessments as part of the study every 3 months during the study period: total bile acids, bile acid profile, fibroblast growth factor 19, and 7-alpha-C4
  Participants will undergo gadoxate-enhanced magnetic resonance imaging at baseline, 12 months, and 36 months.
  Interventions: Drug: Fenofibrate (drug); Diagnostic Test: Blood draw for the laboratory assessment; Diagnostic Test: MRI using a hepatobiliary phase contrast agent (Gd-EOB-DPTA)
- Historical control (No Intervention): Historical control of individuals who underwent liver transplantation for primary sclerosing cholangitis who were not treated with any peroxisome proliferator activated receptor agonist treatment.

INTERVENTIONS:
Drug: Fenofibrate (drug) — Once daily fenofibrate for 36 months
  Arms: Treatment
Diagnostic Test: Blood draw for the laboratory assessment — Serum assessments will be performed every 3 months during the study period
  Arms: Treatment
Diagnostic Test: MRI using a hepatobiliary phase contrast agent (Gd-EOB-DPTA) — Participants will undergo a quantitative gadoxetate-enhanced MRI and MRCP at baseline, and at 12 months and 36 months of trial participation.
  Arms: Treatment

SUMMARY:
This study aims to determine the efficacy of 36 months once-daily fenofibrate in preventing clinically-detectable recurrence of primary sclerosing cholangitis after liver transplantation, compared with a historical control cohort that was not treated with

DETAILED DESCRIPTION:
Primary sclerosing cholangitis (PSC), an immune-mediated, progressive cholestatic disease with no well-established pharmacologic treatment, has an annual incidence of 2.0 per 100,000 and is responsible for 5% of liver transplants (LT) performed in the United States. Recurrent PSC (rPSC) after LT occurs in 8-27% at 5 years and is associated with an over 40% risk of graft loss.

Because PSC patients undergo LT at a younger age than non-PSC patients (median 40-50 years vs 60 years for most other LT indications), rPSC poses significant lifetime morbidity and mortality risk, and development of its early signs of biliary injury, particularly the development cholestasis (elevated alkaline phosphatase), is routinely monitored in the post-transplant setting.

There is no established pharmacologic treatment for rPSC, and the disease is usually characterized by progressive cholestasis to biliary stricturing, cholangitis, allograft fibrosis and ultimately liver failure. Trials of ursodeoxycholic acid and oral vancomycin have been inconclusive. Since most transplants for PSC are performed with Roux-en-Y biliary reconstructions that make re-transplantation challenging, any pharmacologic intervention to reduce the risk of rPSC would represent a breakthrough in disease management.

Cholestasis appears to be a surrogate for PSC disease progression since improvement in alkaline phosphatase levels is associated with slower disease progression, lower rates of cholangiocarcinoma, and improved survival in the pre-transplant setting. Peroxisome proliferator-activated receptor (PPAR) agonists (e.g. fenofibrate, bezafibrate, seladelpar, elafibranor) reduce bile acid-mediated biliary injury by downregulating their synthesis and activity, and promoting choleresis. PPAR agonists have demonstrated efficacy in potently improving cholestasis in PSC pre-transplant, and other cholestatic liver diseases post-transplant.

While fibrates have been shown to improve both biochemical and clinical parameters of PSC in non-transplant patients, whether they can prevent clinically detectable rPSC after transplantation has not been studied. Extrapolating the pre-transplant data to the post-transplant setting, this study hypothesizes that mitigating cholestasis with the use of fibrates in transplant recipients may impede the development of rPSC.

In this study, the primary aim is to assess the efficacy of once daily fenofibrate-a well-tolerated, generic PPAR-alpha agonist widely used for dyslipidemia-in preventing clinically detectable rPSC after 36 months of treatment, compared to an untreated control group. (rPSC diagnosis based on established criteria outlined below).

This study also investigates novel serum biomarkers of biliary inflammation may serve as early signals of disease either as an alternative or an adjunct to alkaline phosphatase, and before biliary stricturing occurs. The study will also employ quantitative biliary flow dynamics with gadoxetate-enhanced margentic resonance imaging (MRI) which can identify early biliary strictures, hepatocyte function and onset of fibrosis is being studied as a modality to assess pre-transplant PSC severity.

rPSC diagnosis: The study utilizes established criteria for diagnosis of rPSC, with additional inclusion and exclusion criteria for more stringent rule-out of other post-transplant complications of the biliary tree, as follows.1 The criteria will be applied to patients who are between 1 and 7 years from LT.

* Explant findings consistent with PSC and
* Absence of untreated hepatic arterial thrombosis, stenosis, or other reason for diminished hepatic arterial resistive indices after LT, and
* Absence of ischemic cholangiopathy after LT, defined as the development of biliary strictures within the first year of LT as defined elsewhere32, and
* Absence of untreated biliary anastomotic (post-surgical) stricture, and
* Presence of intrahepatic and/or extrahepatic biliary stricturing characteristic of PSC by magnetic resonance cholangiography, endoscopic retrograde cholangiography, or percutaneous transhepatic cholangiography, and/or
* Liver biopsy with fibrous cholangitis and/or fibro-obliterative lesions with or without ductopenia, consistent with PSC

ELIGIBILITY:
Inclusion criteria:

* Adults aged 18-75 irrespective of gender who have undergone LT for PSC or PSC-related liver malignancy between 1 year and 7 years (inclusive) prior to study enrollment
* Absence of rPSC at time of study enrollment
* At least one of the following additional features that increase risk of rPSC

  * LT performed for cholangiocarcinoma
  * Concurrent inflammatory bowel disease
  * Any episode of cytomegalovirus viremia in the post-transplant period before study enrollment
  * Any episode of acute cellular rejection in the post-transplant period before the study enrollment
* If target enrollment of 40 patients is not achieved during the first 6 months of study, we will remove f(iii) inclusion criteria to expand enrollment to any patient meeting the other inclusion/exclusion criteria.
* Due to lab requirements, we will only enrol patients who are within a 3 hour driving distance of Mayo Clinic Arizona and/or are willing to travel to Mayo Clinic Arizona at 4 month intervals during the study at own cost.

Exclusion criteria:

* Presence of ischemic cholangiopathy which can mimic rPSC
* LT performed for primary biliary cholangitis or autoimmune hepatitis, or PSC with overlapping primary biliary cholangitis or autoimmune hepatitis, which may recur after LT and confound assessment of cholestasis
* Unaddressed post-LT hepatic artery compromise (e.g thrombosis, stenosis) which can mimic rPSC
* History of total colectomy for curative treatment of ulcerative colitis which reduces risk of rPSC
* Baseline GFR <30 ml/min which precludes administration of fenofibrate
* Previously known intolerance or allergy to fenofibrate
* Other clinically significant comorbid condition, including inability to provide consent and psychiatric conditions, which in the opinion of the study team, may interfere with patient treatment, safety, assessment, or compliance with the treatment
* Female participants that are pregnant or planning to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of rPSC in LT recipients treated with fenofibrate, compared with an untreated control cohort. | 36 months
  Proportion of recipients transplanted for PSC who develop rPSC during a 36-month fenofibrate treatment period, compared to the rate of rPSC in a untreated cohort. The diagnosis of rPSC will be made based on established diagnostic criteria (see Study Design)

SECONDARY OUTCOMES:
To quantify the associations between serum alkaline phosphatase and rPSC development in LT recipients treated with fenofibrate | 36 months
  Quantify the relative risk between serum alkaline phosphatase level (IU/L) and the diagnosis of rPSC (based on established diagnostic criteria - see Study Design) at 36 months of fenofibrate treatment
To quantify the associations between total serum bile acid level and rPSC development in LT recipients treated with fenofibrate | 36 months
  Quantify the relative risk between total serum bile acid level (micromol/liter) with a diagnosis of rPSC (based on established diagnostic criteria - see Study Design) at 36 months of treatment
To quantify the associations between serum bile acid profile and rPSC development in LT recipients treated with fenofibrate | 36 months
  Quantify the relative risk between primary bile acids level (nanonmol/mL), secondary bile acid level (nanonmol/mL), and glycine:taurine conjugate bile acid level (nanonmol/mL) with a diagnosis of rPSC (based on established diagnostic criteria - see Study Design) at 36 months of fenofibrate treatment
To quantify the associations between fibroblast growth factor 19 level and rPSC development in LT recipients treated with fenofibrate | 36 months
  Quantify the relative risk between serum fibroblast growth factor 19 level (picogram/ml) with a diagnosis of rPSC (based on established diagnostic criteria - see Study Design) at 36 months of treatment
To quantify the associations between serum 7-alpha-hydroxy-4-cholesten-3-one level and rPSC development in LT recipients treated with fenofibrate | 36 months
  Quantify the relative risk between serum 7-alpha-hydroxy-4-cholesten-3-one (7-alpha-C4) (nanogram/mL) levels with a diagnosis of rPSC (based on established diagnostic criteria - see Study Design) at 36 months of treatment
To quantify the association between quantitative biliary flow dynamics demonstrated by gadoxetate-enhanced and T1 mapping magnetic resonance imaging with rPSC development in LT recipients treated with fenofibrate | 36 months
  The ANALI score, biliary transit time, and relative enhancement index of the hepatic parenchyma will be quantified by gadoxetate-enhanced MRI/MRCP. These measures will be correlated with the development of rPSC (based on established diagnostic criteria - see Study Design) during fenofibrate treatment period at 12 months, and 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Channa Jayasekera, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials